CLINICAL TRIAL: NCT04685967
Title: Clinical Evaluation of a Restorative Glass Ionomer and a Bulk-fill Composite Resin
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Dr. Fatma Dilşad Öz, Assoc. Prof., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: glass ionomer-bulk fill
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Tooth Disease
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glass-ionomer (Experimental): Equia Forte HT, GC, Tokyo, Japan (EHT)
  Interventions: Device: Glass ionomer
- Bulk-Fill (Experimental): SonicFill2, Orange, CA, USA (SBF)
  Interventions: Device: Bulk-fill composite

INTERVENTIONS:
Device: Glass ionomer — Equia Forte HT, GC, Tokyo, Japan
  Arms: Glass-ionomer
Device: Bulk-fill composite — SonicFill2, Orange, CA, USA
  Arms: Bulk-Fill

SUMMARY:
The clinical performance of a restorative glass ionomer and bulk-fill resin composite in class II restorations will be evaluated and compared. After recruiting participants with at least 2 approximal caries lesions, all restorations will be placed by a single clinician. All caries lesions will be removed before restoring. Cavities will be divided into two groups: a restorative glass ionomer [Equia Forte HT, GC, Tokyo, Japan (EHT)] and bulk-fill composite resin [SonicFill2, Orange, CA, USA (SBF)] All restorative procedures will be conducted according to manufacturers' instructions. Restorations will be scored using modified United States Public Health Service (USPHS) criteria after a week (baseline) 6, 12, 24, 36 and 48 months. Descriptive statistics will be performed using chi-square tests.

ELIGIBILITY:
Inclusion Criteria:

* age range will be 18 to 65
* patients should have at least 2 approximal caries lesions require restoration
* healthy periodontal status
* a good likelihood of recall availability

Exclusion Criteria:

* poor gingival health
* adverse medical history
* potential behavioral problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Clinical performances of different restorative systems according to USPHS criteria | two years
  Two year results according to USPHS criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No